CLINICAL TRIAL: NCT04292431
Title: Exploration of Variations in Leukocyte Morphological Parameters (MDW and CPD) Using the Beckman Coulter DxH900, Based on the Infectious Condition, Inflammatory State and Response to Corticosteroid Therapy in Septic Patients
Brief Title: Leukocyte MOrphology and CORticosteroids Response in SEPtic Patients (MOCORSEP)
Acronym: MOCORSEP
Status: Completed | Type: Observational
Sponsor: Beckman Coulter, Inc. (Industry)
Collaborators: Hôpital Raymond Poincaré (Other); Saint-Louis Hospital, Paris, France (Other)
Responsible Party: Sponsor
Other Study IDs: MOCORSEP_BEC_2019
Record Dates: First submitted 2020-02-28; First posted 2020-03-03 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Sepsis; Septic Shock; Sepsis Syndrome; Infection
Keywords: Leukocyte morphology; Corticosteroid; MDW; Cell population data; DxH900
MeSH Terms: conditions — Sepsis; Shock, Septic; Systemic Inflammatory Response Syndrome; Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Non-interventional, prospective, monocentric study on the exploration of leukocyte morphological parameters according to the infectious condition and response to corticosteroid therapy of septic patients.

DETAILED DESCRIPTION:
Sepsis is a major public health issue, caused by an organ disorder related to an immune response not controlled by the infection.

Several randomized trials have shown that the combination of glucocorticoids and mineralocorticoids improves the survival rate of patients in septic shock. The optimal use of this therapeutic approach requires identifying the pro-inflammatory phase patients likely to respond to corticosteroid therapy.

Hyperactivation of immune cells is accompanied by morphological changes likely to be characterized by modern hematology instruments, particularly the DxH900 (Beckman Coulter). The DxH900 is able to use specific techniques to determine a significant number of morphological characteristics (CPD or Cell Population Data) for circulating leukocytes. Recently, one of these leukocyte morphological parameters, MDW (Monocyte Distribution Width), has been clinically approved for identifying septic patients or those at risk of developing sepsis. This MDW parameter currently has the CE IVD mark and is approved by the American FDA.

The aim of the study is to explore the hypothesis that leukocyte morphological parameters, including MDW, may constitute functional biomarkers of pro-inflammatory response and help to identify septic patients likely to optimally respond to a combination treatment of glucocorticoids and mineralocorticoids, and thus improve their chances of survival.

The proposed study is a non-interventional, prospective, monocentric cohort study to explore the variation of leukocyte morphological parameters measured on the DxH900 hematology analyzer according to the different infectious conditions of patients ranging from a known or suspected infection to septic shock versus non-infected control patients, and possibly based on the response. This observational cohort study will consist of patients with a known or suspected infection, sepsis or in septic shock on their date of admission into one of the medical or surgical departments and monitored up to day 7 of the hospital stay or on the date of discharge from the hospital, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* an infection (known or suspected)
* sepsis
* sepsis + vasopressor
* septic shock

  * responders to corticosteroid therapy
  * non-responders to corticosteroid therapy

Exclusion Criteria:

* Pregnant women
* Patients with onco-hematological diseases with the presence of blasts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non infected (n=50) Infection (n=50) Sepsis + SOFA > 2 (n=25) Sepsis (SOFA > 2) + vasopressors and lactate ≤ 2 mmol/L (n=25) Septic shock (SOFA > 2 + vasopressor + lactate > 2 mmol/L) (n=25)
Sampling Method: Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Leukocytes morphological parameters differs between patient's groups | 7 days
  The leukocytes morphological parameters determined by DxH900 (CPD and MDW) will be compared between the patient's groups in the cohort:
  * patients with infection
  * patients with sepsis
  * patients with septic shock
  * patients with septic shock responding to corticosteroid treatment
  * patients with septic shock not responding to corticosteroid treatment

SECONDARY OUTCOMES:
Leukocytes morphological parameters preditcs inflammatory status | 7 days
  Identify whether the CPD parameters differ between patients with a pro-inflammatory state for those presenting signs of immunosuppression
Leukocytes morphological parameters preditcs responce to corticosteroids treatments | 7 days
  Explore the relevance of CPD parameters for predicting and monitoring the response to corticosteroid therapy in patients with septic shock.

CONTACTS AND LOCATIONS:
Overall Officials: Djillali Annane, MD, Principal Investigator — Hospital Raymond Poincaré; Pierre Moine, MD, Study Chair — Hospital Raymond Poincaré; Martin Rottman, MD, Study Chair — Hospital Raymond Poincaré; Sylvie Chevret, MD, Study Chair — Hospital Saint Louis Lariboisière Fernand-Widal
Locations (1):
- Hospital Raymond Poincaré, Garches, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Annane D, Renault A, Brun-Buisson C, Megarbane B, Quenot JP, Siami S, Cariou A, Forceville X, Schwebel C, Martin C, Timsit JF, Misset B, Ali Benali M, Colin G, Souweine B, Asehnoune K, Mercier E, Chimot L, Charpentier C, Francois B, Boulain T, Petitpas F, Constantin JM, Dhonneur G, Baudin F, Combes A, Bohe J, Loriferne JF, Amathieu R, Cook F, Slama M, Leroy O, Capellier G, Dargent A, Hissem T, Maxime V, Bellissant E; CRICS-TRIGGERSEP Network. Hydrocortisone plus Fludrocortisone for Adults with Septic Shock. N Engl J Med. 2018 Mar 1;378(9):809-818. doi: 10.1056/NEJMoa1705716. PMID 29490185
- [Background] Annane D, Sebille V, Charpentier C, Bollaert PE, Francois B, Korach JM, Capellier G, Cohen Y, Azoulay E, Troche G, Chaumet-Riffaud P, Bellissant E. Effect of treatment with low doses of hydrocortisone and fludrocortisone on mortality in patients with septic shock. JAMA. 2002 Aug 21;288(7):862-71. doi: 10.1001/jama.288.7.862. PMID 12186604
- [Background] Crouser ED, Parrillo JE, Seymour C, Angus DC, Bicking K, Tejidor L, Magari R, Careaga D, Williams J, Closser DR, Samoszuk M, Herren L, Robart E, Chaves F. Improved Early Detection of Sepsis in the ED With a Novel Monocyte Distribution Width Biomarker. Chest. 2017 Sep;152(3):518-526. doi: 10.1016/j.chest.2017.05.039. Epub 2017 Jun 15. PMID 28625579
- [Background] Crouser ED, Parrillo JE, Seymour CW, Angus DC, Bicking K, Esguerra VG, Peck-Palmer OM, Magari RT, Julian MW, Kleven JM, Raj PJ, Procopio G, Careaga D, Tejidor L. Monocyte Distribution Width: A Novel Indicator of Sepsis-2 and Sepsis-3 in High-Risk Emergency Department Patients. Crit Care Med. 2019 Aug;47(8):1018-1025. doi: 10.1097/CCM.0000000000003799. PMID 31107278